CLINICAL TRIAL: NCT03995654
Title: Research of Burden of Interstititial Lung Diseases in Turkey
Acronym: RBILD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Olcay Ayçiçek, asst. prof., Karadeniz Technical University
Other Study IDs: 2018/176
Record Dates: First submitted 2019-05-30; First posted 2019-06-24 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Lung Diseases, Interstitial; Fibrosis Lung
Keywords: Interstitial Lung Diseases; Fibrotic Lung; Prevalence
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to investigate the etiological distribution of ILD, epidemiological characteristics of ILD cases such as age, gender, geography, smoking, occupation, economic status, education, and comorbidities. Another aim is to make the cost calculation from the first to the diagnosis in the patients diagnosed. Obtaining the missing data related to the ILD of our country is one of our goals.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are not previously diagnosed with ILD will be included in the study.

Exclusion Criteria:

* under 18 years old
* older 80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be a multicenter prospective cross-sectional study in Turkey, that will be the coordinating center of our Department of Chest Diseases
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Etiological distribution | 1 year
  The aim of our study is to investigate the etiological distribution of ILD
Etiological distribution | 1 year
  Geographic distribution of ILD patients according to regions (will be presented as %)
Epidemiological characteristics of ILD cases | 1 year
  Age (years)
Epidemiological characteristics of ILD cases | 1 year
  Gender (male, female; (will be presented as %))
Epidemiological characteristics of ILD cases | 1 year
  Smoking (yes, no; (will be presented as %)
Epidemiological characteristics of ILD cases | 1 year
  Distribution of ILD patients according to the occupation (will be presented as %)
Epidemiological characteristics of ILD cases | 1 year
  Economic status (monthly salary of patients according to ILD types and stages of ILD)
Epidemiological characteristics of ILD cases | 1 year
  Distiribution of ILD patienst according to comorbidities (will be presented as YES or NO and %) Comorbiditites are; Hypertension, Heart failure, Coronary Artery Disease, Arrhythmia, Heart Valve Disease, Asthma, COPD, Chronic Renal Disease, Diabetes Mellitus, Hyper / Hypothyroidism, HIV, Cirrhosis / Chronic Liver Disease, Lung malignancy, Extrapulmonary solid organ malignancy, Hematologic malignancy, SVO, Alzeimer, Epilepsy, Neuromuscular Ill, Organ Transplant Receiver, Reflux, Slyding hernia, Others
Total number | 1 year
  We planned enroll roughly 1000 patients to the study

SECONDARY OUTCOMES:
Clinical findings | 1year
  According to the etiology of ILD, clinical findings (Rod, Ral, Rash, Arthritis, Alopecia, Erythema nodosum, Peripheral lymphadenomegaly, Cyanosis, Edema, Raynaud's phenomenon, Other) will be presented as YES or NO and %
Pulmonary functions | 1year
  According to the etiology of ILD, pulmonary functions, will be assessed; FVC (ml) and (%pred)
Pulmonary functions | 1year
  According to the etiology of ILD, pulmonary functions, will be assessed; FEV 1 (ml) and (%pred)
Pulmonary functions | 1year
  According to the etiology of ILD, pulmonary functions, will be assessed; DLCO (mL.min.mmHg) and (%pred)
Pulmonary functions | 1year
  According to the etiology of ILD, pulmonary functions, will be assessed; DLCO/VA (mL.min.mmHg) and (%pred) 6dk YT (meters) Pulseoksimetre ile PaO2 (%)
Pulmonary functions | 1year
  According to the etiology of ILD, pulmonary functions, will be assessed; 6min Walk Test (meters)
Pulmonary functions | 1year
  According to the etiology of ILD, pulmonary functions, will be assessed; PaO2 with Pulse oximeter (%)
Diagnostic methods | 1year
  According to the etiology of ILD, diagnostic methods used in ILD cases will be presented Diagnoses methods are; Clinical and radiology, Bronchoscopic transbronchial lung biopsy, Bronchoalveolar lavage, Transthoracic needle biopsy with imaging, EBUS, VATS, Thoracotomy, Other (Methods are will be shown as YES or NO and %)
Time | 1year
  According to the etiology of ILD, the time spent for diagnosis will be presented Time will be presented as months.
Treatment methods | 1year
  Determining the treatment preferences of physicians according to the etiology of the cases will be presented; Treatment methods are; Non-treatment monitoring, Symptomatic treatment, Systemic corticosteroid, Cytostatic drugs, Antifibrosan drugs (eg Pirfenidone, Nintedanib), Immunological therapy, Referral to other centers, Preparing for transplantation, Home oxygen therapy, Reflux therapy, Other (Methods are will be shown as YES or NO and %)

CONTACTS AND LOCATIONS:
Locations (1):
- Department Of Chest Diseases, School Of medicine, Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to ethical approve, IPD will not be shared with other researchers unless after ethical approves for any further study, researchers can ask for data